CLINICAL TRIAL: NCT03042013
Title: An Open-label, Multicenter, Rollover Study for Subjects Who Are Participating in an Astellas-sponsored ASP8273 Study
Brief Title: A Study for Subjects Who Are Participating in an Astellas-sponsored ASP8273 Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Following recommendation by SOLAR Study IDMC, Astellas closed enrollment in ASP8273 studies.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8273-CL-0201; 2016-003183-39 (EudraCT Number)
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Subjects With NSCLC With an EGFR Activating Mutation
Keywords: ASP8273; Non-Small-Cell Lung Cancer; EGFR mutations; Oncology
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — naquotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASP8273 (Experimental): Subjects will receive a once or twice daily oral dose of ASP8273 (3 dose strengths)
  Interventions: Drug: ASP8273

INTERVENTIONS:
Drug: ASP8273 — Oral

SUMMARY:
The purpose of the study is to evaluate long-term safety and tolerability of continuous treatment with ASP8273 in subjects who are participating in an Astellas-sponsored ASP8273 study which has completed, at a minimum, the primary analysis or have completed the individual study evaluation period and for whom the investigator feels the subject may have potential to continue to derive clinical benefit from treatment with ASP8273.

DETAILED DESCRIPTION:
This is a multicenter, rollover study for subjects with non-small cell lung cancer (NSCLC) with an epidermal growth factor receptor (EGFR) activating mutation who are currently participating in studies evaluating ASP8273.

Subjects should sign the informed consent at cycle 1 day 1 visit. The assessments from the last treatment visit from the parent study can be utilized for the cycle 1 day 1 visit. Either local or central laboratories may be utilized for the cycle 1 day 1 visit if assessments are used from the last treatment visit of the parent study. The subject will then receive ASP8273 study drug for the rollover study and return all ASP8273 study drug from the parent study. Subjects will continue on to subsequent 28-day cycles until 1 of the discontinuation criteria are met. Upon enrollment, subjects with fewer than 6 cycles of study drug dosing in the parent study will return to the clinic on day 1 of each cycle up to cycle 5. After cycle 5, these subjects can switch to day 1 of every other odd cycle for clinic visits. Subjects with 6 or more cycles of study drug dosing upon enrollment into the rollover study will return to the clinic on day 1 of every other odd cycle (e.g., cycles 3, 5, etc.). Imaging methods and frequency will be performed per standard of care.

An end of treatment study visit will be conducted 30 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be participating in an Astellas-sponsored ASP8273 study which has completed, at a minimum, the primary analysis or have completed the individual study evaluation period requirements. Subject must not have met any discontinuation criteria in the parent study.
* Subject must be receiving a stable dose of ASP8273 for 14 days minimum and is able to enroll into this rollover study without treatment interruption of study drug, or with no more than 21 consecutive days of treatment interruption in study drug within the parent study.
* Subject should be deriving clinical benefit without any persistent intolerable toxicity from continued treatment of ASP8273.
* Subject agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Subject who developed persistent intolerable toxicity to ASP8273 treatment in the parent study.
* Subject who received any other systemic anticancer treatment after parent study entry (radiation to local areas such as bone or brain if received in the parent ASP8273 study is permitted).
* Subject who requires the following medications will be excluded:

  * Chemotherapy, radiotherapy, immunotherapy or other medications intended for antitumor activity
  * Investigational products or therapy other than ASP8273
  * Strong inhibitors or inducers of CYP3A4
  * Permeability-glycoprotein (P-gp) substrates with a narrow therapeutic index
* Subject has any condition which may require treatment during the study and may make the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (safety and tolerability) | Up to a maximum of 1 month (per cycle)
  An Adverse Event (AE) is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product
Number of participants with laboratory value abnormalities and/or adverse events related to treatment | Up to a maximum of 1 month (per cycle)
  Number of participants with potentially clinically significant laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.

IPD SHARING:
Plan to Share IPD: Undecided